CLINICAL TRIAL: NCT04662242
Title: The Prognostic Impact of Selenium On Critical Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201902287A3A0
Record Dates: First submitted 2020-11-29; First posted 2020-12-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Critical Illness; Selenium Deficiency; Trace Element Deficiency; Acute Abdomen; Sepsis
MeSH Terms: conditions — Critical Illness; Abdomen, Acute; Sepsis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low serum selenium with selenium supplement (Experimental): Patients having low serum selenium with selenium supplement given
  Interventions: Drug: Selenium Supplement
- low serum selenium with placebo supplement (Placebo Comparator): Patients having low serum selenium with placebo given
  Interventions: Drug: normal saline
- non-low serum selenium with selenium supplement (Active Comparator): Patients having normal serum selenium with selenium supplement given
  Interventions: Drug: Selenium Supplement
- non-low serum selenium with placebo supplement (Placebo Comparator): Patients having normal serum selenium with placebo given
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Selenium Supplement — Zelnite 400mcg/day in normal saline 100ml iv infusion for 7 days
  Other Names: Zelnite
  Arms: low serum selenium with selenium supplement; non-low serum selenium with selenium supplement
Drug: normal saline — normal saline 100ml iv infusion for 7 days
  Arms: low serum selenium with placebo supplement; non-low serum selenium with placebo supplement

SUMMARY:
Selenium is an important trace element for human for its multiple roles such as the antioxidant activity. Previous evidences showed that critically ill patients may benefit from selenium supplement but the dose and results are controversial.

Patients after operations for acute abdomen usually suffer from sepsis and stress. The aim of this study is to investigate the efficacy of selenium replacement in critical patients of acute abdomen, to see the impact on prognosis.

DETAILED DESCRIPTION:
Acute abdomen is a common surgical emergency and is often the result of peritonitis due to an acute inflammatory process within abdominal cavity. Many of the patients with acute abdomen have severe sepsis and are critically ill that require an emergency surgery.

The mortality rate of such patients are high because these patients usually have a profound pathophysiological dysregulation and multiple organ dysfunction. One of the mechanism of is the loss of anti-oxidative capacity of cells that fail to recover from ischemic-reperfusion injury.

Selenium is an important cofactor that participate in the antioxidant activity of glutathione peroxidase reaction. There are evidences that critically ill patients may benefit from selenium supplement by better outcome and less mortality but the dose and results are still heterogenous and inconclusive.

The aim of this study is to investigate the efficacy of selenium replacement in critical patients of acute abdomen, to see if there is a significant impact on prognosis, and to establish a clinical guide in the future.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit (ICU) patients receiving abdominal surgeries for acute abdomen
* within 48 hours post-operatively
* stay in ICU for more than 48 hours
* meets sepsis criteria of Sepsis-3 (2016)

Exclusion Criteria:

* liver cirrhosis Child-Pugh score B or C
* breastfeeding or pregnancy
* allergy yo selenium
* vegetative status or irreversible diseases with life-expectancy fewer than 28 days
* End-stage renal disease under dialysis
* Human immunodeficiency virus infection
* neutropenia not due to sepsis (granulocyte < 1000/mm3)
* Heart failure (New York Heart Association class III-IV) or recent myocardial infarction (within 6 weeks)
* post cardiopulmonary cerebral resuscitation within 4 weeks
* taking immunosuppressants
* receiving anti-cancer therapy
* signed do not resuscitation
* joined other clinical research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
mortality rate | 30 day
  mortality rate in 30 days

SECONDARY OUTCOMES:
hospital length | 1 year
  hospital length for current admission
ventilator length | 1 year
  ventilator length for current admission
complication rate | 30 days
  complication rate within 30 days
organ failure rate | 30 days
  organ failure rate within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Tung Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] Allingstrup M, Afshari A. Selenium supplementation for critically ill adults. Cochrane Database Syst Rev. 2015 Jul 27;2015(7):CD003703. doi: 10.1002/14651858.CD003703.pub3. PMID 26214143